CLINICAL TRIAL: NCT04590625
Title: Apatinib Mesylate Combined With Albumin Binds Paclitaxel and Carboplatin or Cisplatinum as First-line Treatment for Stage II-IV Epithelial Ovarian Cancer Followed by Apatinib Maintenance Therapy:a Single-arm,Exploratory Clinical Study
Brief Title: Apatinib Combined With Abraxane and Carboplatin or Cisplatinum as First-line Treatment for Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-O001
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib; Albumin-Bound Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): 1. Neoadjuvant therapy:
     Apatinib:apatinib one course will last 21 days.Oral administration at a dose of 250 mg, qd; Abraxane:abraxane one course will last 21 days.Intravenously guttae at a dose of 260 mg/m2,d1; Cis-platinum or Carboplatin:cis-platinum or carboplatin one course will last 21 days.cis-platinum introperitoneal injection at a dose of 75-100 mg/m2,d1;carboplatin intravenous injection at a dose of AUC=5-6,d1.
     Neoadjuvant therapy is 3-4 cycles.After Neoadjuvant therapy will received interval cytoreductive surgery.
  2. Adjuvant therapy:
     After interval cytoreductive surgery,patients will received adjuvant therapy same as neoadjuvant therapy.
     Adjuvant therapy is 3 cycles
  3. maintenance treatment: After above treatment finished,patients will received aptinib for 2 years.
  Interventions: Drug: Apatinib Mesylate; Drug: Abraxane; Drug: Cis Platinum; Drug: Carboplatin
- Group2 (Experimental): 1.Adjuvant therapy:
  After primary cytoreductive surgery,patients will received adjuvant therapy:
  Apatinib:apatinib one course will last 21 days.Oral administration at a dose of 250 mg, qd; Abraxane:abraxane one course will last 21 days.Intravenously guttae at a dose of 260 mg/m2,d1; Cis-platinum or Carboplatin:cis-platinum or carboplatin one course will last 21 days.cis-platinum introperitoneal injection at a dose of 75-100 mg/m2,d1;carboplatin intravenous injection at a dose of AUC=5-6,d1.
  Adjuvant therapy is 3 cycles 3.maintenance treatment: After above treatment finished,patients will received aptinib for 2 years.
  Interventions: Drug: Apatinib Mesylate; Drug: Abraxane; Drug: Cis Platinum; Drug: Carboplatin

INTERVENTIONS:
Drug: Apatinib Mesylate — apatinib one course will last 21 days.Oral administration at a dose of 250 mg, qd
Drug: Abraxane — abraxane one course will last 21 days.Intravenously guttae at a dose of 260 mg/m2,d1
Drug: Cis Platinum — cis-platinum one course will last 21 days.cis-platinum introperitoneal injection at a dose of 75-100 mg/m2,d1
Drug: Carboplatin — carboplatin one course will last 21 days.carboplatin intravenous injection at a dose of AUC=5-6,d1

SUMMARY:
This monocentric, prospective, observational study will evaluate the safety and efficacy of apatinib in combination with albumin binds paclitaxel and carboplatin or cisplatinum as first-line treatment for stage II-IV epithelial ovarian cancer followed by apatinib maintenance therapy in routine clinical practice. Eligible patients will be followed for approximately 20 months.

ELIGIBILITY:
Inclusion Criteria:

-

1.Age 18 - 75 years; 2.Histologically confirmed, stage II or IV epithelial ovarian carcinoma; 3.For Group1,patients with stage III-IV ovarian cancer who are considered unlikely to achieve satisfactory tumor reduction after preoperative evaluation by gynecological oncologists or not suitable for direct surgery are required; 4.Patients with at least one evaluable or measurable lesions as per RECIST version 1.1(CT scan length and diameter of tumor lesion≥10mm CT scan of lymph node lesion was short diameter≥15mm,scan slice thickness 5mm); 5.ECOG performance status (PS) 0 - 2; 6.Life expectancy of at least 12 weeks; 7.Patients with adequate organ function at the time of enrollment as defined below:

1. Blood routine examination standard:(without blood transfusion within 14 days before enrollment)

   1. Hb ≥ 100g/L，
   2. WBC ≥ 3.0×109/L
   3. ANC ≥ 1.5×109/L，
   4. PLT ≥ 100×109/L；
2. Biochemical examination shall meet the following standards:

   1. BIL ≤ 1.5 times the upper limit of normal(ULN);
   2. ALT and AST ≤ 3 ×upper limit of normal(ULN);
   3. Serum creatinine Cr ≤ 1ULN;
   4. Serum creatinine ALB ≥ 30g/L. 8.Women of childbearing age in the serum or urine pregnancy test is negative within 7 days prior to study enrollment and must be Non-lactating patients,and agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 8 months after the end of the study; males should agree to patients who must use contraception during the study period and within 8 months after the end of the study period.

      9.Subjects voluntarily joined the study, signed informed consent, good compliance, and followed up;

      Exclusion Criteria:
      1. Women who are pregnant or breastfeedind;
      2. Except for other malignant tumors, basal cell carcinoma of the skin and cervical cancer in situ in the past 5 years;
      3. Patients with symptomatic brain metastasis;Significant neurological or psychiatric disorders;
      4. Patients who have participated in other clinical trials in recent three months;
      5. Prior treatment with apatinib or other anti-vascular drugs and other small molecule tyrosine kinase inhibitors;
      6. Patients who have undergone systemic chemotherapy, radiotherapy, surgery, hormone therapy, or immunotherapy before enrollment;
      7. Within 3 months before treatment, there were esophageal (gastric fundus) varicose bleeding, intestinal obstruction and gastrointestinal perforation;
      8. Patients had clinically demonstrated cancerous ascites or pleural effusion;
      9. Patients has active infection or unexplained fever ≥38.5℃ within 7 days before enrollment;
      10. Severe liver, kidney, heart, lung, brain and other major organ failure;
      11. Patients with hypertension that is difficult to control (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents;
      12. Previous or current had idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, histopathological pneumonia (e.g., bronchitis, obliterans), drug-induced pneumonia, or screening stage CT with active pneumonia;
      13. Patients with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds), bleeding tendency or receiving thrombolytic or anticoagulant therapy are allowed to receive low-dose LMWH or oral aspirin to prevent anticoagulant therapy during the trial;
      14. Urine protein ≥ ++ or confirmed 24 hour urine protein quantitation;
      15. Patients with cardiac clinical symptoms or diseases that are not well controlled,such as:(1) NYHA2 or above heart failure;(2) Unstable angina;(3) Myocardial infarction occurred within 1 year;(4) Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention;(5) QTc > 470ms;
      16. Inability to swallow pills, malabsorption syndrome, or any condition that affects gastrointestinal absorption;
      17. In the 6 months prior to enrollment, patients had been arteriovenous thrombosis (AVT), such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis (DVT) and pulmonary embolism;
      18. Patients with a history of hereditary or acquired bleeding or coagulation disorders.There were clinically significant bleeding symptoms or definite bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding and hemorrhagic gastric ulcer;
      19. According to the judgment of the researcher, the patients have other factors that may lead to the forced termination of this study, such as other serious diseases (including mental diseases) requiring combined treatment, severe laboratory test abnormalities, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | approximately 2 years
  defined as the proportion of patients with no gross tumor tissue residual after interval cytoreductive surgery
Progression-free survival | approximately 2 years
  defined as time from first administration of first-line therapy to documented disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiao, Doctor, Principal Investigator — Zhongshan Hospital Xiamen University
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No